CLINICAL TRIAL: NCT05138302
Title: A Prospective Multicenter Clinical Study of BRCA and DNA Damage Repair Genes in Blood Samples of Chinese Pancreatic Cancer Patients
Brief Title: A Clinical Study of BRCA and DNA Damage Repair Genes in Blood Samples of Chinese Pancreatic Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CPOG2021015
Record Dates: First submitted 2021-10-27; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — This study is an observe research

SUMMARY:
This study aims to know the status of BRCA and DDR genes in PDAC patients in China. Peripheral venous blood samples of the patients will be collected for next-generation sequencing of BRCA and DNA damage repair related genes. At the same time, it is necessary to record clinical information such as age, gender, tumor pathological type, tumor stage and grade, whether surgery is performed, the size of postoperative residual lesions, and treatment methods. Prognostic indicators include the association of factors such as PFS, ORR, and DCR are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pancreatic cancer
* PS score ≤ 2
* no severe heart, cerebrovascular disease, severe coagulation dysfunction or severe mental disorder

Exclusion Criteria:

* PS score > 2
* with severe heart, cerebrovascular disease, severe coagulation dysfunction or severe mental disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with pancreatic cancer
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-04-19 (Estimated); Study Completion 2023-04-19 (Estimated)

PRIMARY OUTCOMES:
OS | 2years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- RenJiH, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided